CLINICAL TRIAL: NCT05027997
Title: Exploratory Phase 2a Randomized, Double-blind, Placebo-controlled Study of Dipraglurant (ADX48621) Immediate Release Tablets in Patients With Blepharospasm
Brief Title: Exploratory Study of Dipraglurant (ADX48621) for the Treatment of Patients With Blepharospasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Addex Pharma S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADX48621-203
Record Dates: First submitted 2021-07-29; First posted 2021-08-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2021-11

CONDITIONS: Blepharospasm; Dystonia
Keywords: Blepharospasm; Dystonia
MeSH Terms: conditions — Blepharospasm; Dystonia | interventions — 6-fluoro-2-(4-(pyridin-2-yl)but-3-yn-1-yl)imidazo(1,2-a)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dipraglurant 50 mg (Experimental)
  Interventions: Drug: Dipraglurant
- Dipraglurant 100 mg (Experimental)
  Interventions: Drug: Dipraglurant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dipraglurant — Oral tablet
  Other Names: ADX48621
  Arms: Dipraglurant 100 mg; Dipraglurant 50 mg
Drug: Placebo — Oral matching placebo tablet
  Arms: Placebo

SUMMARY:
This study is designed to assess the safety and tolerability of dipraglurant in patients with blepharospasm (BSP) (randomized 1:1:1 to receive dipraglurant 50 mg, 100 mg or placebo) and explore the efficacy of 50 mg and 100 mg immediate release tablets (versus placebo) on the severity and frequency of BSP signs and symptoms using objective measures, clinical ratings and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of idiopathic benign essential blepharospasm
* Must have had prior response to to botulinum toxin (BoNT) reported on last 2 consecutive injection cycles
* Last injection of BoNT at least 8 weeks prior to Screening assessments
* Patient is experiencing features of Blepharospasm (BSP) of moderate severity/frequency at study entry.

Exclusion Criteria:

* BSP that is known or suspected to be associated with a known cause such as neuroleptic exposure, brain injury or lesion, stroke, Parkinson's disease, or related Parkinsonisms
* History of surgical intervention (e.g., deep brain stimulation) or orbital myectomy for dystonia
* Disabling eyelid opening apraxia
* Other neurological disease (including psychiatric disease and/or cognitive impairment) that, in the opinion of the investigator, would affect the patient's ability to complete study assessments.
* Other significant medical condition that may affect the safety of the patient or preclude adequate participation in the study.

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of dipraglurant as measured by incidence of adverse events | Baseline to Day 2
  The primary outcome will be testing the safety and tolerability of dipraglurant in patients with blepharospasm based on the incidence of adverse events reported by patients and/or as identified by the Investigator based on clinical assessments conducted during the study.
Computerized Motor Objective Rater (CMOR) analysis of blinking activity | Baseline to Day 2
  Video analysis, by an independent rater, of the mean proportion of eye closure time, severity of periocular spasms, and blink rate. Decreased eye closure time, severity of periocular spasms and blink rate indicates improvement of blepharospasm symptoms.
Skintronics wearable analysis of blinking activity | Baseline to Day 2
  Analysis of blinking activity as recorded on the Skintronics wearable device. Decreased blink activity indicates improvement of blepharospasm symptoms.

SECONDARY OUTCOMES:
Jankovic Rating Scale (JRS) severity score | Baseline to Day 2
  The JRS is a clinician rated scale for blepharospasm. The intensity of eyelid spasms is measured based on a 5 point grading system where 0 indicates no symptoms and 4 indicates the most severe symptoms.
Jankovic Rating Scale (JRS) frequency score | Baseline to Day 2
  The JRS is a clinician rated scale for blepharospasm. The frequency of eyelid spasms is measured based on a 5 point grading system where 0 indicates no symptoms and 4 indicates highest frequency symptoms.
Global Dystonia Severity Rating Scale (GDS) | Baseline to Day 2
  The GDS is a clinician rated scale for the assessment of dystonia severity across multiple body regions. Each body region is rated on a scale from 0-10 where 0 represents no dystonia and 10 represents severe dystonia.
Blepharospasm Phenotyping Tool (BPT) | Baseline to Day 2
  The BPT is a clinician rated scale assessing 4 major phenotypic elements of blepharospasm using a 4 point scale for severity and frequency, where 0 indicates no symptoms and 4 indicates the highest frequency and/or most severe symptoms.
Blepharospasm Severity Rating Scale (BSRS) | Baseline to Day 2
  The BSRS is a clinician rated scale for rating severity of blepharospasm based on 6 clinical features of the condition. A total score is generated based on the combined score for severity and frequency and where a higher value indicates more severe symptoms.
Clinician's Global Impression of Severity (CGI-S) score | Baseline to Day 2
  The CGI-S score is used by the Investigator to determine, in a global sense, how severe the patients blepharospasm is in the context of other blepharospasm patients. Increased scores indicate more severe symptoms.
Blepharospasm Disability Index (BSDI) | Baseline to Day 2
  The BSDI is a 6 item patient rated disability scale that measures how blepharospasm effects activities of daily living. Each item is scored on a 5 point scale to produce a total score of up to 30, where a higher individual item score and a higher total score indicate greater disability to the patient.
Patient Global Impression of Change (PGI-C) score | Baseline to Day 2
  The PGI-C score is a patient reported outcome that assesses how much the blepharospasm symptoms have improved or worsened. A score of 0 indicates no change, negative scores down to -3 indicate worsening, and positive scores of up to 3 indicate improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No